CLINICAL TRIAL: NCT03825380
Title: Efficacy and Safety Assessment of T4032 Versus Lumigan® in Ocular Hypertensive or Glaucomatous Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LT4032-301
Record Dates: First submitted 2019-01-21; First posted 2019-01-31 (Actual); Results first posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-02

CONDITIONS: Ocular Hypertension; Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma | interventions — Bimatoprost

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T4032 (Experimental)
  Interventions: Drug: Bimatoprost
- Lumigan® (Active Comparator)
  Interventions: Drug: Lumigan®

INTERVENTIONS:
Drug: Bimatoprost — Eyedrops
  Arms: T4032
Drug: Lumigan® — Eyedrops
  Arms: Lumigan®

SUMMARY:
The purpose of this study is to assess the efficacy and safety of T4032 versus Lumigan.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed and dated.
* Both eyes with diagnosed open-angle glaucoma or ocular hypertension

Exclusion Criteria:

* History of trauma, infection, clinically significant inflammation within the 3 previous months.
* Uncontrolled diabetic patient.
* Pregnancy or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2018-11-23 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-02-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital, Tallinn, Estonia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 485 patients (from 723 screened patients) were included and randomised in the study: 485 patients in the intent-to-treat (ITT) set and Safety set, 469 in the modified ITT (mITT) set.
  The recruitment started on 23-NOV-2018 and was completed on 28-AUG-2020 and the last patient completed the study on 24-FEB-2021.
Pre-assignment Details: Incl/Excl criteria checked at screening visit, then patients discontinued their current treatment to start the run-in period with Azopt, for 5 weeks. The Azopt was stopped 1 or 2 weeks before the randomisation visit (Day 1). Incl/Excl criteria are confirmed at Day 1. 723 screened patients, 485 randomised patients, 238 screen failure patients.
Period: Overall Study
Arm/Group | T4032 | Lumigan®
Started | 236 | 249
Completed | 218 | 227
Not Completed | 18 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T4032 | Lumigan® | Total
Number analyzed (Participants) | 236 | 249 | 485
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 126 | 125 | 251
  >=65 years | 110 | 124 | 234
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.03 (11.85) | 63.67 (10.92) | 63.36 (11.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 153 | 294
  Male | 95 | 96 | 191
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Estonia | 6 | 8 | 14
  Belgium | 5 | 3 | 8
  Bulgaria | 41 | 39 | 80
  Canada | 4 | 3 | 7
  Czechia | 21 | 19 | 40
  France | 10 | 13 | 23
  Georgia | 5 | 7 | 12
  Germany | 4 | 4 | 8
  Greece | 4 | 9 | 13
  Hungary | 2 | 0 | 2
  Italy | 13 | 12 | 25
  Latvia | 9 | 11 | 20
  Lithuania | 4 | 3 | 7
  Mauritius | 1 | 0 | 1
  Poland | 20 | 27 | 47
  Russia | 30 | 31 | 61
  Slovakia | 10 | 12 | 22
  Spain | 14 | 14 | 28
  Tunisia | 17 | 19 | 36
  Ukraine | 16 | 14 | 30
  United Kingdom | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Intra-Ocular Pressure
Description: Change from Baseline to Week 12 in Intra Ocular Pressure in mmHg in the worse eye
Time Frame: Week 12
Population: Modified Intent To Treat
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | T4032 | Lumigan®
Number analyzed (Participants) | 229 | 240
mmHg | -9.67 (0.19) | -9.50 (0.18)
Statistical Analysis 1: Comparison: T4032 vs Lumigan®; Test type: Non-Inferiority — Primary tested:Non-inferiority of T4032 to Lumigan® on the change from baseline in IOP using a MMRM. 3 independent models will be performed, one for each time point (8:00, 10:00 & 16:00). The 95% CI for treatment effect (difference T4032 - Lumigan) will be estimated at Wk 12. NI will be achieved if the upper bound of the 95% CI for the difference between treatment groups (T4032 - Lumigan) is lower than the margin of +1.5 mmHg for each of the 3 time points 8:00, 10:00 & 16:00; p = 0.453, Mixed Models Analysis; Adjusted Mean Difference = -0.17, 95% CI 2-sided [-0.62 to 0.28], Standard Error of Mean 0.23

ADVERSE EVENTS:
Time Frame: Adverse event reporting extends from start of the treatment until Day 112 follow-up phone call.
Arm/Group | T4032 | Lumigan®
All-Cause Mortality (participants affected / at risk) | 0/236 | 0/249
Serious Adverse Events (participants affected / at risk) | 1/236 | 2/249
Other Adverse Events (participants affected / at risk) | 13/236 | 17/249
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T4032 (N=236) | Lumigan® (N=249)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T4032 (N=236) | Lumigan® (N=249)
Conjunctival hyperaemia (Eye disorders) | 13 (13) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the results of the Trial are the sole and exclusive property of THEA, and cannot be used in whatever form without prior written agreement of THEA.

DOCUMENTS (2):
  • Study Protocol (2019-07-05): https://cdn.clinicaltrials.gov/large-docs/80/NCT03825380/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT03825380/SAP_001.pdf